CLINICAL TRIAL: NCT00107861
Title: A Phase I/II Study of Interferon-Beta Gene Transfer (Ad.hIFN-β) in the Treatment of Refractory Colorectal Carcinoma With Liver Metastases
Brief Title: Interferon-Beta Gene Transfer (Ad.hIFN-β) as Treatment for Refractory Colorectal Carcinoma With Liver Metastases
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Study MD
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201-20
Record Dates: First submitted 2005-04-11; First posted 2005-04-12 (Estimated); Last update posted 2009-07-14 (Estimated); Status verified 2009-07

CONDITIONS: Colorectal Carcinoma; Metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis

INTERVENTIONS:
Drug: Ad.hIFN-β (BG00001, IDEC-201)

SUMMARY:
This study will be conducted in subjects with refractory colorectal carcinoma with unresectable liver metastases. The purposes of the study are:

* to evaluate the safety and any harmful effects of an intravenous injection of Ad.hIFN-β;
* help determine whether the virus carrying the interferon-beta gene will enter the bloodstream and liver tumor cells and cause the cancer cells to die.

DETAILED DESCRIPTION:
This trial is a clinical research study of Ad.hIFN-β, an investigational, replication-defective, recombinant adenovirus containing the human interferon beta gene, for people that have refractory colorectal carcinoma with liver metastases. Scientists have been exploring a variety of approaches to develop medications to treat patients with refractory colorectal carcinoma with liver metastases; a disease for which current treatment provides only limited relief, so there is a need for new medications.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically confirmed hepatic metastases from primary colorectal carcinoma.
* Not amenable to complete surgical resection for attempted cure as determined by the Principal Investigator (PI).
* Tumor progression after prior therapy for colorectal carcinoma, including fluoropyrimidine (5 FU or capecitabine), irinotecan, oxaliplatin, or cetuximab.
* One or more metastatic hepatic tumors that is measurable on CT scan. In addition, subjects may have nonhepatic metastatic tumors.
* ECOG performance status of ≤ 1.
* Age ≥ 18 years.
* Signed, written IRB-approved informed consent.
* Men and women of reproductive potential must be willing to follow accepted birth control methods during treatment and for 3 months after completion of treatment.
* Acceptable liver function:

  * Bilirubin ≤ 1.5 x upper limit of normal;
  * AST, ALT ≤ 2.0 x upper limit of normal;
  * Albumin ≤ 3.0 g/dL.
* Acceptable hematologic status:

  * Granulocyte ≥ 1000 cells/mm3;
  * Platelet count ≥ 150,000 plts/mm3;
  * Hemoglobin > 9 g/dL.
* Acceptable coagulation status: INR within normal limits.
* Acceptable kidney function: Serum creatinine within normal limits.

Exclusion Criteria:

* New York Heart Association Class III or IV cardiac disease, myocardial infarction within the past 6 months prior to Day 1, unstable arrhythmia, or evidence of ischemia on ECG within 14 days prior to Day 1.
* Seizure disorders requiring anticonvulsant therapy.
* Severe chronic obstructive pulmonary disease with hypoxemia.
* Major surgery, other than diagnostic surgery, within 4 weeks prior to Day 1.
* Active uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy.
* Pregnant or nursing women.
* Treatment with radiation therapy, surgery, chemotherapy, or investigational therapy within 1 month prior to study entry.
* Unwillingness or inability to comply with procedures required in this protocol.
* Known infection with HIV, hepatitis B, or hepatitis C.
* Serious nonmalignant disease (e.g., hydronephrosis, liver failure, or other conditions) that could compromise protocol objectives in the opinion of the investigator and/or the sponsor.
* Clinically significant bleeding event within the last 3 months, unrelated to trauma.
* More than 50% of liver replaced by tumor (estimated by the PI from CT scan within 14 days of Day 1).
* Previous treatment with Ad.hIFN-β.
* Any prior treatment with a gene delivery vector or an adenovirus therapeutic agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44
Dates: Start 2005-05; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
- Evaluate the safety of a single IV administration of Ad.hIFN-β.

SECONDARY OUTCOMES:
Evaluate the MTD or maximum feasible dose (MFD) of Ad.hIFN-β.
Evaluate IFN-β and Ad.hIFN-β vector serum concentrations.
Evaluate immunogenicity of Ad.hIFN-β by measuring human anti adenovirus and human anti-IFN-β antibody formation.
Explore preliminary clinical activity.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of California San Diego, La Jolla, California
  - Mary Crowley Medical Research Center, Dallas, Texas